CLINICAL TRIAL: NCT04859049
Title: Assessing the Effect of Single Injection Infromedial Peribulbar Injection in Lacrimal Duct Intubation Surgery in Adult Patient: Prospective Cohort Study
Brief Title: Single Injection Infromedial Peribulbar Injection in Lacrimal Duct
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Research Institute of Ophthalmology, Egypt (Other)
Responsible Party: Principal Investigator, Abeer Samir Salem, Researcher of anesthesia, Research Institute of Ophthalmology, Egypt
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: anesth RIO
Record Dates: First submitted 2021-04-04; First posted 2021-04-26 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Pain Due to Certain Specified Procedures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental): Infra- medial injection of local anesthesia mixture
  Interventions: Procedure: infromedial single injection
- Group 2 (Experimental): medial canthus injection of the local anesthesia mixture
  Interventions: Procedure: medial canthus injection

INTERVENTIONS:
Procedure: infromedial single injection — Group 1: We used a 25G/ 1" length needle to inject 3ml of lidocaine: bupivacaine (1:1) with 30 IU hyaluronic acid, 0.5ml below the inferior punctum in the lower lid medial margin.
  Arms: Group 1
Procedure: medial canthus injection — : We used a 25G/ 1" length needle to inject 3ml of lidocaine: bupivacaine (1:1) with 30 IU hyaluronic acid classical medial canthal injection
  Arms: Group 2

SUMMARY:
infromedial injection of 3 ml local anesthetic drugs and assessing the pain during lacrimal duct intubation and probability of false tracking

DETAILED DESCRIPTION:
After entering the OR; the patient will be cannulated and fully monitored with basic monitors (pulse oximeter, NIBP & ECG), a nasal cannula is connected to the patient to deliver oxygen.

We gave the patient 5 ml of propofol to decrease the discomfort felt by the patient during injection of local anesthesia. Benox eye drops is applied to the operative eye in both groups.

Patients were allocated into 2 groups; each group is 25 patients Group 1: We used a 25G/ 1" length needle to inject 3ml of lidocaine: bupivacaine (1:1) with 30 IU hyaluronic acid, 0.5ml below the inferior punctum in the lower lid medial margin.

Group 2: We used a 25G/ 1" length needle to inject 3ml of lidocaine: bupivacaine (1:1) with 30 IU hyaluronic acid classical medial canthal injection

During surgery, we will assess the pain degree during probing using Verbal Rating Scale (0 to 10 scale where 0 is no pain an 10 is unbearable pain), to assess the efficiency of this single low volume injection.

ELIGIBILITY:
Inclusion Criteria:

* adults undergoing lacrimal duct intubation surgery
* Patients' physical status by the American Association of Anesthesiology (ASA): ASA I, II, III.
* Age between 18-70, both sexes.
* Axial lengths ranging between 22-28mm.

Exclusion Criteria:

* ASA IV.
* Patient age less than 18 or more than 70 years.
* Coagulation disorders (e.g. patients on warfarin (INR<1.5)
* Communication difficulties preventing reliable assessment.
* High myopia (axial length more than 28mm) and medial staphylomas.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-09-10 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Verbal rating scale (VRS) is a 5 point scale from 0 to 4 where 0 is no pain and 4 is unbearable pain | during surgery , study will started September 2021 & will end November 2022
  pain scale

SECONDARY OUTCOMES:
surgery satisfaction using yes or no questionnaire | during surgery
  easiness and false tracking of the dilators

CONTACTS AND LOCATIONS:
Overall Officials: abeer salem, MD, Principal Investigator — research institute of ophthalmology
Locations (2):
- Egypt (2):
  - Research Institute of Ophthamology, Giza
  - Research Institute of Ophthalmology, Giza

IPD SHARING:
Plan to Share IPD: No